CLINICAL TRIAL: NCT02480816
Title: Cardiometabolic Response to a Sodium-bicarbonated Mineral Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, M Pilar Vaquero, Scientific researcher, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BW-13
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Mineral Waters

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Bicarbonated mineral water (BW) (Experimental): Bicarbonated mineral water
  Interventions: Dietary Supplement: Mineral water
- Control mineral water (CW) (Active Comparator): Mineral water low in mineral content (control)
  Interventions: Dietary Supplement: Mineral water

INTERVENTIONS:
Dietary Supplement: Mineral water — Intake of 1 L per day of the mineral water (BW or CW) with main meals, crossover design

SUMMARY:
The effects of consuming a sodium-bicarbonated mineral water rich in bicarbonate, sodium, chloride, lithium and silicon are studied in humans. The aim of this assay was to determine whether the consumption of this water as part of the usual diet, reduces cardiometabolic risk factors in adult men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, men and women >18 and ≤ 45 years
* Total-cholesterol > 200 mg/dL and < 300 mg/dL

Exclusion Criteria:

* Age <18 and > 45 years
* Total-cholesterol ≥300 mg/dL
* Triglycerides > 250 mg/dL
* Total-cholesterol / HDL-cholesterol > 6
* Being a usual consumer of carbonic mineral water
* BMI < 20 and >30 kg/m2
* Diabetes
* Hypertension or digestive, liver or renal disease
* Eating disorders
* Being under medication that could affect lipid metabolism
* Consumption of functional foods that could affect lipid metabolism (food containing n-3 fatty acids or phytosterols)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | Baseline
LDL-cholesterol | 4 weeks
LDL-cholesterol | 8 weeks

SECONDARY OUTCOMES:
Total-cholesterol | Baseline
Total-cholesterol | 4 weeks
Total-cholesterol | 8 weeks
Triglycerides | Baseline
Triglycerides | 4 weeks
Triglycerides | 8 weeks
HDL-cholesterol | Baseline
HDL-cholesterol | 4 weeks
HDL-cholesterol | 8 weeks
Apolipoprotein A | Baseline
Apolipoprotein A | 4 weeks
Apolipoprotein A | 8 weeks
Apolipoprotein B | Baseline
Apolipoprotein B | 4 weeks
Apolipoprotein B | 8 weeks
Glucose | Baseline
Glucose | 4 weeks
Glucose | 8 weeks
Insulin | Baseline
Insulin | 4 weeks
Insulin | 8 weeks
Urine creatinin | Baseline
Urine creatinin | 8 weeks
Urine calcium | Baseline
Urine calcium | 8 weeks
Urine potassium | Baseline
Urine potassium | 8 weeks
Urine sodium | Baseline
Urine sodium | 8 weeks
Urine pH | Baseline
Urine pH | 8 weeks
Systolic Blood Pressure | Baseline
Systolic Blood Pressure | 4 weeks
Systolic Blood Pressure | 8 weeks
Diastolic Blood Pressure | Baseline
Diastolic Blood Pressure | 4 weeks
Diastolic Blood Pressure | 8 weeks
Oxidized LDL | Baseline
Oxidized LDL | 4 weeks
Oxidized LDL | 8 weeks
Serum aldosterone | Baseline
Serum aldosterone | 8 weeks
BMI | Baseline
BMI | 4 weeks
BMI | 8 weeks
Dietary energy intake | Baseline
Dietary energy intake | 8 weeks
Dietary protein intake | Baseline
Dietary protein intake | 8 weeks
Dietary fat intake | Baseline
Dietary fat intake | 8 weeks
Dietary cholesterol intake | Baseline
Dietary cholesterol intake | 8 weeks
Dietary carbohydrate intake | Baseline
Dietary carbohydrate intake | 8 weeks

REFERENCES:
- [Result] Toxqui L, Vaquero MP. An Intervention with Mineral Water Decreases Cardiometabolic Risk Biomarkers. A Crossover, Randomised, Controlled Trial with Two Mineral Waters in Moderately Hypercholesterolaemic Adults. Nutrients. 2016 Jun 28;8(7):400. doi: 10.3390/nu8070400. PMID 27367723